CLINICAL TRIAL: NCT06167187
Title: Is Inferior Alveolar Nerve Block Beneficial in Fracture Mandibular Surgeries? A Randomised Controlled Trial
Brief Title: The Effect of Inferior Alveolar Nerve Block in Fracture Mandibular Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, mohamed atef, assistant lecturer of anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MD94/2023
Record Dates: First submitted 2023-12-02; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Anesthesia
MeSH Terms: interventions — Ketorolac; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (IAN block group) (Active Comparator): patients will receive bilateral inferior alveolar nerve block. 23 patients
  Interventions: Procedure: bilateral inferior alveolar nerve block
- control group (Active Comparator): patients will not receive the block and will receive intravenous multimodal analgesia according to standard protocol.
  23 patients
  Interventions: Drug: Ketorolac and fentanyl

INTERVENTIONS:
Procedure: bilateral inferior alveolar nerve block — Placing the tip of the thumb or forefinger into the coronoid notch (retromolar fossa) to help visualize the vertical height at which the needle will enter, and retracting the cheek to expose the pterygomandibular triangle. Placing the barrel of the syringe over the contralateral lower 1st and 2nd premolars and resting the side of the needle tip against the lateral edge of the pterygomandibular raphe, aiming the tip of the needle into the pterygomandibular triangle, with the bevel facing the ramus. Advancing the needle tip slightly into the mucosa until it is stopped by the ramus (typically after about 2 to 2.5 cm of insertion) and withdrawing needle 1 mm away from bone. Aspirating to rule out intravascular placement. If aspiration reveals intravascular placement, withdrawal of the needle will be done 2 to 3 mm, then reaspirating prior to injection. Slowly injecting about 2 to 4 milliliters of bupivacaine 0.5% anesthetic in each side..
  Other Names: IANB
  Arms: Study group (IAN block group)
Drug: Ketorolac and fentanyl — in control group, Patients will not receive the block and pain will be controlled according to institutional protocol using 30 mg ketorolac IV and fentanyl increments as needed.
  Arms: control group

SUMMARY:
The aim of the study is to assess the efficacy of adding of pre-emptive inferior alveolar nerve block compared to the conventional systemic intravenous analgesia in controlling perioperative pain in fracture mandibular surgeries.

DETAILED DESCRIPTION:
Opioid drug administration is a common technique to reduce pain from surgical trauma. However, the use of large doses of opioid drugs during and after surgery can be associated with an increased incidence of multiple side effects such as; ventilatory depression, sedation, nausea, vomiting, pruritus, difficult voiding and ileus.

In maxillofacial surgeries in which patients often receive maxillomandibular fixation these side effects are troublesome to the patient and at worst case scenario can cause a life-threatening complications. Ventilatory depression and vomiting are the most serious side effects especially in early postoperative hours. Various methods have been proposed to minimize these side effects. Nerve block with long-acting local anesthesia is a proposed technique in this regard.

In maxillofacial operations, bupivacaine is a highly efficient long-acting local anesthetic and has been used as a safe local anesthetic for neuroanalgesia after cleft lip operation or third molar surgery alone or in combination with low-power laser and diclofenac.

Inferior alveolar nerve block is considered as gold standard for sensory block of the hemi mandible. It can provide adequate anesthesia and analgesia for one side of the mandibular teeth and gingival mucosa, the body and inferior ramus of the mandible, the anterior two-thirds of the tongue and floor of the mouth cavity.

The inferior alveolar nerve (IAN) block is a widely used regional anaesthetic nerve block for the mandible. The most commonly used technique for IAN block is called the direct approach which include inserting the needle into the pterygomandibular raphae by penetrating the buccinators muscle. Once in this space, the aim is to inject the local anaesthetic solution besides the inferior alveolar nerve before it enters the mandibular foramen.

ELIGIBILITY:
Inclusion Criteria:

1. Age group: 18 - 65 years old.
2. American Society of Anesthesiologists (ASA) Physical Status Class I to III
3. Scheduled for fracture mandible fixation.

Exclusion Criteria:

1. Refusing to participate in the study.
2. History of allergy to the medications used in the study.
3. Contraindications to regional anesthesia (including coagulopathy and local infection).
4. Psychiatric disorders.
5. Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
The time of the first dose of fentanyl rescue analgesia intraoperative | Throughout the surgery
  guided by hemodynamic changes
Total amount of additional intraoperative fentanyl rescue analgesia | Throughout the surgery
  guided by hemodynamic changes
The time from recovery to the first dose pethidine rescue analgesic | 24 hours postoperatively
  guided by visual analogue scale.
Total amount of pethidine postoperative rescue analgesic | 24 hours postoperatively
  guided by visual analogue scale.

SECONDARY OUTCOMES:
Incidence of complications related to the block | 24 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Atef, ass.lecturer, Principal Investigator — faculty of medicine, ain shams university
Locations (1):
- Faculty of medicine - Ain shams university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No